CLINICAL TRIAL: NCT06500715
Title: Acupuncture as add-on to GCS-F Treatment for Reducing Febrile Neutropenia-related Hospitalization in Patients Undergoing Doxorubicin-based Treatment for Sarcoma: a Randomized Crossover Study
Brief Title: Acupuncture as add-on to G-CSF for Febrile Neutropenia-related Hospitalization in Doxorubicin-treated Patients With Sarcoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Noah Samuels, Director, Center for Integrative Complementary Medicine, Shaare Zedek Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ACP-CIFN.2024
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Febrile Neutropenia; Sarcoma; Doxorubicin Adverse Reaction; Hospitalization-Associated Infection
Keywords: febrile neutropenia; acupuncture; sarcoma; doxorubicin; hospitalization
MeSH Terms: conditions — Febrile Neutropenia; Sarcoma; Cross Infection | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Participating patients will be treated with one of the following doxorubicin-based protocols, for between 4 and 6 cycles: Doxorubicin and Dacarbazine (AD regimen); Doxorubicin and Ifosfamide (AI regimen); or Doxorubicin and Cisplatin (AC regimen). Subcutaneous 6mg of pegylated G-CSF (pegfilgrastim-jmdb, Fulphila) will be administered at 24h following chemotherapy.
  Allocation to study groups: Study patients will be randomly allocated (1:1) to one of the two study treatment arms: Group A, undergoing the acupuncture intervention at the 1st chemotherapy cycle; no acupuncture at the 2nd cycle; intervention at the 3rd; and so on. Group B: No intervention at the 1st cycle; acupuncture intervention at the 2nd cycle; and so on. T
Who Masked: Care Provider
Masking Description: he treating oncologist will be blinded as to the patient's allocation and study intervention during each cycle of chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Patients in Group A will undergo the acupuncture intervention at the 1st chemotherapy cycle; no acupuncture at the 2nd cycle; intervention at the 3rd; and so on.
  Interventions: Device: Acupuncture
- Group B (Active Comparator): No intervention at the 1st cycle; acupuncture intervention at the 2nd cycle; and so on.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Acupuncture will be administered bilaterally on points PC6, LI 4, CV6, SP6, SP10 and ST36 on the first day of each cycle (d1), prior to administration of chemotherapy; and on d8, each session lasting between 30 to 45 minutes. Patients will continue from d1 to d8 with press-tack acupuncture needles on points PC 6, LI4, SP 6 and ST 36. On d8, patients will again undergo acupuncture, and continue with self-acupressure on the same points as the press-tack needles, until the next chemotherapy cycle.
  Other Names: Acupuncture needle; Press-Tack needle; Self-Acupressure

SUMMARY:
Chemotherapy-induced febrile neutropenia (CIFN) is a dangerous complication of many chemotherapy drugs, with current treatment with granulocyte colony-stimulating factors (G-CSFs) accompanied by adverse effects, primarily muscle and bone pain. Adult patients with sarcoma treated with doxorubicin-based chemotherapy have a high risk (>40%) for developing CIFN. Acupuncture has been shown to have a potentially myelo-protective effect on bone marrow during chemotherapy, though its effect on the incidence of CIFN-related hospitalization has yet to be examined. In the proposed study, patients with sarcoma will be randomly allocated (in a ratio of 1:1) to Group A, receiving acupuncture during cycles 1, 3, and 5; or Group B, during cycles 2, 4, and 6, with the study oncologist blinded regarding allocation. Acupuncture will be administered on the first day (d1) and the 8th day (d8) of the chemotherapy cycles, with press-tack needles on d1 to d8, and patients will be taught to self-treat with acupressure from d8 to the next cycle. The incidence and duration of hospitalization due to CIFN will be examined, as will adherence to the chemotherapy regimen; G-CSF-related pain; and other outcomes using 3 quality-of-life-focused questionnaires. The study findings will have important implications regarding the role of acupuncture in the treatment of patients treated with chemotherapy drugs with a high risk for CIFN, such as those used in the treatment of sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* diagnosed with sarcoma of any stage
* scheduled for doxorubicin-based chemotherapy
* function ECOG status score of 0-1

Exclusion Criteria:

* not fulfilling all inclusion criteria
* unwilling or unable to provide written informed consent for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of chemotherapy-induced febrile neutropenia-related hospitalization | 3 weeks
Duration of chemotherapy-induced febrile neutropenia-related hospitalization | 3 weeks

SECONDARY OUTCOMES:
Relative Dose Intensity of Chemotherapy Regimen | 3 weeks
  Actual vs. planned dosage and interval between cycles
G-CSF-related muscle and bone pain | 3 wseks
  Patient-reported outcome measures
Quality of life-related outcomes: Quantitative Assessment | 3 weeks
  Patient-reported outcome measures
Quality of life-related outcomes: Qualitative Assessment | 3 weeks
  MYCaW narratives
Adverse effects of study intervention | 3 weeks
  Patient medical files

CONTACTS AND LOCATIONS:
Overall Officials: Noah Samuels, MD, Principal Investigator — Shaare Zeded Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyman GH, Bohlke K, Cohen L. Integrative Therapies During and After Breast Cancer Treatment: ASCO Endorsement of the SIO Clinical Practice Guideline Summary. J Oncol Pract. 2018 Aug;14(8):495-499. doi: 10.1200/JOP.18.00283. No abstract available. PMID 30096271
- [Background] Mao JJ, Ismaila N, Bao T, Barton D, Ben-Arye E, Garland EL, Greenlee H, Leblanc T, Lee RT, Lopez AM, Loprinzi C, Lyman GH, MacLeod J, Master VA, Ramchandran K, Wagner LI, Walker EM, Bruner DW, Witt CM, Bruera E. Integrative Medicine for Pain Management in Oncology: Society for Integrative Oncology-ASCO Guideline. J Clin Oncol. 2022 Dec 1;40(34):3998-4024. doi: 10.1200/JCO.22.01357. Epub 2022 Sep 19. PMID 36122322
- [Background] Shih YW, Su JY, Kung YS, Lin YH, To Anh DT, Ridwan ES, Tsai HT. Effectiveness of Acupuncture in Relieving Chemotherapy-induced Leukopenia in Patients With Breast Cancer: A Systematic Review With A Meta-Analysis and Trial Sequential Analysis. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211063884. doi: 10.1177/15347354211063884. PMID 34930039
- [Background] Nian J, Sun X, Zhao W, Wang X. Efficacy and safety of acupuncture for chemotherapy-induced leukopenia: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Oct 21;101(42):e30995. doi: 10.1097/MD.0000000000030995. PMID 36281119
- [Background] Li S, Huang J, Guo Y, Wang J, Lu S, Wang B, Gong Y, Qin S, Zhao S, Wang S, Liu Y, Fang Y, Guo Y, Xu Z, Ulloa L. PAC1 Receptor Mediates Electroacupuncture-Induced Neuro and Immune Protection During Cisplatin Chemotherapy. Front Immunol. 2021 Sep 6;12:714244. doi: 10.3389/fimmu.2021.714244. eCollection 2021. PMID 34552585
- [Background] Samuels N, Ben-Arye E. Integrative Medicine for Cancer-Related Pain: A Narrative Review. Healthcare (Basel). 2024 Feb 4;12(3):403. doi: 10.3390/healthcare12030403. PMID 38338288